CLINICAL TRIAL: NCT03534596
Title: Surgery for Adhesive Small Bowel Obstruction in a Defined Population: a Cohort Study
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: ASBO-01
Record Dates: First submitted 2018-05-10; First posted 2018-05-23 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Adhesive Small Bowel Obstruction
Keywords: cohort; surgery; adhesive small bowel obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cohort study of patients operated for adhesive small bowel obstruction (SBO) during a five-year period

DETAILED DESCRIPTION:
It is a population-based cohort study of patients operated for adhesive small bowel obstruction during a five-year period (2007-2012) in two Swedish neighboring regions. Patients were identified by a broad search of operation and ICD codes. Preoperative data as age, gender, co-morbidity, previous surgery was registered as well as mechanisms of obstruction and intraoperative data. Short and long-term complications were analyzed. Patients were followed to 31st January 2017 , last medical note or death.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Surgery for adhesive small bowel obstructions during the time period 2007-2011 in Uppsala County and Gävle County, Sweden

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery due to adhesive small bowel obstructions during the time period 2007 -2011.
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of surgery for SBO | 1st January 2007 - 31st December 2011
  per 100 000 inhabitants and year

SECONDARY OUTCOMES:
Short term surgical complications | From surgery until <30 days postoperatively
  anastomotic leaks, intraabdominal abscesses, wound dehiscence, wound infection, urinary tract infection, cardiopulmonary events, use of antibiotics, re-operation, ICU-care, death
Long term surgical complications | >30 days postoperatively until death or 31st of January, 2017
  re-admissions for SBO, re-operations for SBO, hernias and mortality
Relationships between complications and pre- and intraoperative variables | From surgery until death or 31st of January, 2017

CONTACTS AND LOCATIONS:
Overall Officials: Urban Karlbom, MD PhD, Study Chair — Region Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sakari T, Christersson M, Karlbom U. Mechanisms of adhesive small bowel obstruction and outcome of surgery; a population-based study. BMC Surg. 2020 Apr 6;20(1):62. doi: 10.1186/s12893-020-00724-9. PMID 32252752